CLINICAL TRIAL: NCT05462873
Title: A Phase I/Ib, Open-label, Multi-center, Study of QEQ278 in Patients With Advanced Solid Tumors
Brief Title: A Study to Investigate the Safety and Tolerability of Intravenous QEQ278 in Patients With Advanced Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CQEQ278A12101
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck
Keywords: NKG2D; NKG2D-L; immunotherapy; ADCC; NK cells; NSCLC; ESCC; RCC; HPV-associated HNSCC; QEQ278
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma, Renal Cell; Esophageal Squamous Cell Carcinoma; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose escalation (Experimental): Dose escalation with QEQ278 single agent
  Interventions: Biological: QEQ278
- Part 2: Dose expansion (Experimental): Dose expansion with QEQ278 single agent
  Interventions: Biological: QEQ278

INTERVENTIONS:
Biological: QEQ278 — Intravenous dosing of QEQ278

SUMMARY:
To characterize safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary anti-tumor activity of QEQ278 in adult patients with advanced/metastatic non-small cell lung cancer, esophageal squamous cell carcinoma, renal cell carcinoma, and human papilloma virus associated head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
This study is an open-label, phase I/Ib, multi-center study of QEQ278 as a single agent, consisting of a dose escalation part followed by a dose expansion part.

In the dose escalation part of the study, patients with non-small cell lung cancer (NSCLC), esophageal squamous cell carcinoma (ESCC), renal cell carcinoma (RCC), or human papilloma virus (HPV)-associated head and neck squamous cell carcinoma (HNSCC) will be treated with QEQ278 single agent until the maximum tolerated dose (MTD) is reached or a lower recommended dose (RD) is established.

The study may enter the dose expansion, after an MTD(s) and/or RD(s) is declared in the dose escalation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent must be obtained prior to participation in the study.
* Adult men and women ≥ 18 years of age.
* Histologically confirmed and documented advanced malignancies (locally advanced malignancies, non-curable by surgery or radiotherapy and metastatic disease). Disease must be measurable, including presence of at least one measurable lesion, as determined by RECIST v1.1.
* In the opinion of the treating investigator, patients must have received, but are not benefitting from standard therapies, be intolerant or ineligible to receive such therapy, or have no standard therapy option for the respective disease types (diseases listed below), as well as any other therapies deemed to be standard by local/institutional standard.
* Non-small cell lung cancer
* Esophageal squamous cell carcinoma
* Renal cell carcinoma
* HPV-associated head and neck squamous cell carcinoma
* Must have a site of disease amenable to biopsy and be a candidate for tumor biopsy according to the treating institution's guidelines. The patient must be willing to undergo a new tumor biopsy at screening and during treatment.

Exclusion Criteria:

* Active previously documented or suspected autoimmune disease. Patients with vitiligo, type I diabetes, residual hypothyroidism only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur should not be excluded. Patients previously exposed to anti-PD-1/PD-L1 treatment who are adequately treated for skin rash or with replacement therapy for endocrinopathies should not be excluded.
* Patients with a history of or current interstitial lung disease or pneumonitis ≥ Grade 2.
* Patients who discontinued prior anti-PD-1 therapy due to an anti-PD-1-related toxicity
* Clinically significant cardiac disease or risk factors at screening
* Insufficient bone marrow function at screening:
* Infections:
* Known history of testing positive for Human Immunodeficiency Virus infection.
* Active Hepatitis B and / or Hepatitis C.
* Active, documented COVID-19 infection
* Known history of tuberculosis
* Any serious uncontrolled infection (acute or chronic).
* Systemic chronic steroid therapy (>10 mg/day prednisone or equivalent) or any immunosuppressive therapy, other than replacement-dose steroids in the setting of adrenal insufficiency, within 7 days of the first dose of study treatment. Topical, inhaled, and ophthalmic steroids are allowed.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-04-04 (Actual); Primary Completion 2026-01-20 (Estimated); Study Completion 2026-01-20 (Estimated)

PRIMARY OUTCOMES:
Incidence and nature of Dose Limiting Toxicities (DLTs) during the DLT evaluation period for single agent QEQ278 | 28 days
  A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the DLT evaluation period and meets the criteria defined in the study protocol.
Incidence and severity of adverse events (AEs) and serious adverse events (SAEs) | Up to 31 months
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs), including changes in laboratory values, vital signs, and electrocardiograms (ECGs) qualifying and reported as AEs.
Frequency of dose interruptions, reductions | Up to 30 months
  Number of dose interruptions of QEQ278 and number of dose reductions of QEQ278
Dose intensity | Up to 30 months
  Dose intensity of QEQ278 is defined as the ratio of actual cumulative dose received and actual duration of exposure.

SECONDARY OUTCOMES:
Overall response rate (ORR) per RECIST v1.1 | Up to 30 months
  ORR is defined as the proportion of patients with a confirmed BOR of complete response (CR) or partial response (PR) by local investigator review as per RECIST v1.1.
Disease control rate (DCR) per RECIST v1.1 | Up to 30 months
  DCR is defined as the proportion of patients with a confirmed best overall response (BOR) of CR or PR or stable disease (SD) by local investigator review as per RECIST v1.1.
Duration of Response (DOR) per RECIST v1.1 | Up to 30 months
  DOR is defined as the time form the date of the first documented response (CR or PR) to the date of the first documented progression by local investigator review as per RECIST v1.1 or death due to underlying cancer.
Progression-free survival (PFS) per RECIST v 1.1 | Up to 30 months
  PFS is defined as the time from the date of start of treatment to the date of the first documented progression by local investigator review as per RECIST v1.1, or death due to any cause.
Peak serum concentration (Cmax) of QEQ278 | During first 168 days of treatment
  The maximum (peak) serum drug concentration after single dose administration
Area under the concentration time curve (AUC) last of QEQ278 | During first 168 days of treatment
  The AUC from time zero to the last measurable concentration sampling time
Area under the concentration time curve (AUC) infinity of QEQ278 | During first 168 days of treatment
  The AUC from time zero to infinity
Time to reach peak serum concentration (Tmax) of QEQ278 | During first 168 days of treatment
  The time to reach maximum (peak) serum drug concentration after single dose administration
Elimination half-life (T1/2) of QEQ278 | During first 168 days of treatment
  The elimination half-life associated with the terminal slope of a semi logarithmic concentration-time curve
Total body clearance (CL) of QEQ278 | During first 168 days of treatment
  The total body clearance of drug from the serum
Volume of distribution (Vz) of QEQ278 | During first 168 days of treatment
  The apparent volume of distribution during terminal phase
Incidence of anti-drug antibody (ADA) | Day 1 and 15
  Immunogenicity of QEQ278

CONTACTS AND LOCATIONS:
Locations (12):
- United States (4):
  - University of California LA, Los Angeles, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Massachusetts General Hospital Dept. of Mass General Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
- Novartis Investigative Site, Brussels, Belgium
- Novartis Investigative Site, Paris, France
- Novartis Investigative Site, Essen, Germany
- Novartis Investigative Site, Milan, MI, Italy
- Novartis Investigative Site, Kashiwa, Chiba, Japan
- Novartis Investigative Site, Singapore, Singapore
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- Novartis Investigative Site, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No